CLINICAL TRIAL: NCT01999348
Title: A Study of GANFORT® UD in Patients With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT) in a Medical Setting
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/039
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma, Primary Open Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Timolol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with POAG or OHT: Patients with POAG or OHT treated with GANFORT® UD (fixed combination bimatoprost and timolol) administered in accordance with physician standard practice for up to 12 weeks.
  Interventions: Drug: Fixed Combination Bimatoprost and Timolol

INTERVENTIONS:
Drug: Fixed Combination Bimatoprost and Timolol — Patients with POAG or OHT treated with GANFORT® UD (fixed combination bimatoprost and timolol) administered in accordance with physician standard practice for up to 12 weeks.
  Other Names: GANFORT® UD

SUMMARY:
The study will evaluate patients diagnosed with POAG or OHT who are switched to GANFORT® UD (unit dose of fixed combination bimatoprost and timolol) therapy for medical reasons in accordance with physician standard clinical practice. All treatment decisions lie with the physician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma or ocular hypertension
* Previously prescribed intraocular pressure (IOP)-lowering medication with insufficient IOP control and is now being switched to GANFORT® UD for medical reasons

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary open-angle glaucoma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1553 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2014-12-19 (Actual); Study Completion 2014-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Wiesloch, Germany

REFERENCES:
- [Background] Pfennigsdorf S, Eschstruth P, Hasemeyer S, Feuerhake C, Brief G, Grobeiu I, Shirlaw A. Preservative-free bimatoprost 0.03%/timolol 0.5% fixed combination in patients with glaucoma in clinical practice. Clin Ophthalmol. 2016 Sep 20;10:1837-1846. doi: 10.2147/OPTH.S106159. eCollection 2016. PMID 27703324

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With POAG or OHT
Started | 1553
Completed | 1433
Not Completed | 120

BASELINE CHARACTERISTICS:
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1553
Age, Customized [Number; unit: participants]
  Less than 18 years | 1
  18 to 30 years | 8
  31 to 40 years | 21
  41 to 50 years | 119
  51 to 60 years | 313
  61 to 70 years | 415
  71 to 80 years | 477
  81 to 90 years | 155
  Greater than or equal to 91 | 8
  Missing data | 36
Sex/Gender, Customized [Number; unit: participants]
  Female | 913
  Male | 631
  Missing data | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) in the Study Eye
Description: IOP is a measure of the fluid pressure inside the study eye. A result at the Final Visit that is lower than the result at Baseline indicates a reduction in IOP (improvement).
Time Frame: Baseline, Final Visit (Week 8 to 12)
Population: Participants from the Per-protocol population, all treated participants who had no major protocol violations, with complete data available at Baseline and Final Visit for analyses.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1321
mmHg
  Baseline | 22.18 (3.55)
  Final Visit | 16.11 (2.87)

2. Secondary Outcome: Physician Assessment of IOP-Lowering Effect in the Study Eye Using a 3-Point Scale
Description: The physician assessed the effectiveness of Ganfort® UD with regard to IOP changes from Baseline using a 3-point scale where: 1=Better than expected (best), 2=As expected and 3=Worse than expected. The number of participants in each category is reported.
Time Frame: Baseline, Final Visit (Week 8 to 12)
Population: Per-protocol population included all treated participants who had no major protocol violations.
Measure: Number; unit: participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1391
participants
  Better than expected | 497
  As expected | 729
  Worse than expected | 98
  Missing data | 67

3. Secondary Outcome: Patient Assessment of Tolerability on a 4-Point Scale
Description: The patient assessed the tolerability of Ganfort® UD using a 4-point scale where: 1=very good (best), 2=good, 3=moderate and 4=poor. The number of participants in each category is reported.
Time Frame: Final Visit (Week 8 to 12)
Population: Per-protocol population included all treated participants who had no major protocol violations.
Measure: Number; unit: participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1391
participants
  Very good | 788
  Good | 461
  Moderate | 45
  Poor | 50
  Missing | 47

4. Secondary Outcome: Physician Assessment of Tolerability on a 4-Point Scale
Description: The physician assessed the patient's tolerability of Ganfort® UD using a 4-point scale where: 1=very good (best), 2=good, 3=moderate and 4=poor. The number of participants in each category is reported.
Time Frame: Final Visit (Week 8 to 12)
Population: Per-protocol population included all treated participants who had no major protocol violations.
Measure: Number; unit: participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1391
participants
  Very good | 809
  Good | 474
  Moderate | 40
  Poor | 28
  Missing | 40

5. Secondary Outcome: Percentage of Patients Who Discontinued Treatment
Description: The percentage of participants who discontinued treatment with Ganfort® UD up to the Week 12 Final Visit
Time Frame: 12 Weeks
Population: Per-protocol population included all treated participants who had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1391
percentage of participants | 6.47

6. Secondary Outcome: Percentage of Patients Prescribed by the Physician to Continue Treatment
Description: The percentage of participants who continued treatment with Ganfort® UD after Week 12.
Time Frame: Final Visit (Week 8 to 12)
Population: Per-protocol population included all treated participants who had no major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1391
percentage of participants | 89.14

7. Secondary Outcome: Physician Assessment of Patient Compliance Compared to Previous Treatment on a 3-Point Scale
Description: The physician assessed patient compliance with Ganfort® UD compared to previous treatment using a 3-point scale where: 1=better (best), 2=equal and 3=worse. The number of participants in each category is reported.
Time Frame: Final Visit (Week 8 to 12)
Population: All participants from the Per-protocol population, all treated participants who had no major protocol violations, who received previous treatment.
Measure: Number; unit: participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1352
participants
  Better | 727
  Equal | 542
  Worse | 34
  Missing | 49

ADVERSE EVENTS:
Time Frame: Up to 12 Weeks
Description: Participating physicians were required to document all serious adverse events (SAEs), irrespective of relationship, and all non-serious adverse drug reactions (ADRs).
Arm/Group | Patients With POAG or OHT
Serious Adverse Events (participants affected / at risk) | 1/1553
Other Adverse Events (participants affected / at risk) | 0/1553
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With POAG or OHT (N=1553)
Death (General disorders) | 1 — The patient died at the age of 78 years. According to the attending ophthalmologist, no further information regarding cause of death was available. The physician assessed the causal relation between the fatal outcome and Ganfort® UD as 'unrelated'.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.